CLINICAL TRIAL: NCT06654999
Title: A Precision Study To Demonstrate The Repeatability and Reproducability of DERM Outputs
Brief Title: How Consistent is the Output of DERM, When Used to Assess Images of Potentially Cancerous Skin Lesions.
Status: Completed | Type: Observational
Sponsor: Skin Analytics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: DERM-011
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Skin Cancer; Melanoma of Skin; Squamous Cell Cancer; Basal Cell Cancer
Keywords: Precision; DERM; Repeatability; Reproducability
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Neoplasms, Squamous Cell; Neoplasms, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients: All patients will have their skin lesion imaged in the same way
  Interventions: Device: Deep Ensemble for the Recognition of Malignancy (DERM)

INTERVENTIONS:
Device: Deep Ensemble for the Recognition of Malignancy (DERM) — DERM variants "+" and "DS"

SUMMARY:
DERM is a Medical Device that uses artificial intelligence to help doctors check if a skin lesion might be cancerous. It works by analysing close-up pictures of skin lesions taken with a smartphone.

This study aims to demonstrate how consistent (precise) the output of DERM is: i.e. does it provide the same result when it analyses multiple photos of the same lesion (repeatability), and when the same lesion is photographed by different people, or with different cameras (reproducibility).

Adults with at least one skin lesion that doctors are checking for cancer, as part of their standard care, will be able to take part. Suitable lesions will be photographed three times, each by three different people using three sets of image capture hardware (specifically, an iPhone 11 with a DL200/HR dermoscopic lens). Each image will be checked for good image quality as it is captured. Images will then be transferred to DERM, where they'll be analysed.

The DERM output won't be shared with the patients or doctors involved in the study. The patients will continue to have their skin lesion biopsy/excised, in accordance with standard of care. Their diagnosis will be collected and compared to the output from DERM.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female,
* aged 18 years or above,
* Willing and able to give informed consent for participation in the study,
* Has at least one skin lesion that, following assessment by a primary care provider and a dermatology specialist, will be biopsied due to a high suspicion of skin cancer, and is suitable for assessment by DERM.
* In the Investigator's opinion, able and willing to comply with all study requirements.

Exclusion Criteria:

* Patients with more than one skin lesion due for biopsy
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

To be suitable for inclusion, a skin lesion must NOT have ANY of the following limitations:

* Be located on an anatomical site of different skin structure: palms of hands or soles of feet (acral lesion), mucosal surfaces (lips and eyes) or under nail (ungal lesion),
* Have a diameter greater than the diameter of the dermoscopic lens,
* Be located on an anatomical site unsuitable for photographing, including on surface of genitals and hair-bearing areas,
* Have been previously biopsied, excised, treated or is otherwise traumatised
* Be located in an area of visible scarring or tattooing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in specialist dermatology clinics in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Reproducibility: Average Positive Agreement (APA) of DERM on malignant lesions is >80% | 1 day
  Each lesion will be imaged by three users using three sets of the image capture hardware, generating nine data sets (user/hardware combinations) per lesion. Each lesion image data set will consist of 3 repeated measures, resulting in 27 measures per lesion
Repeatability: Average Positive Agreement (APA) of DERM on malignant lesions is >80% | 1 day
  Each lesion will be imaged by three users using three sets of the image capture hardware, generating nine data sets (user/hardware combinations) per lesion. Each lesion image data set will consist of 3 repeated measures, resulting in 27 measures per lesion.

SECONDARY OUTCOMES:
Reproducibility: Average Negative Agreement (ANA) of DERM on benign lesions is >50% | 1 day
  Each lesion will be imaged by three users using three sets of the image capture hardware, generating nine data sets (user/hardware combinations) per lesion. Each lesion image data set will consist of 3 repeated measures, resulting in 27 measures per lesion.
Repeatability: Average Negative Agreement (ANA) of DERM on benign lesions is >50% | 1 day
  Each lesion will be imaged by three users using three sets of the image capture hardware, generating nine data sets (user/hardware combinations) per lesion. Each lesion image data set will consist of 3 repeated measures, resulting in 27 measures per lesion.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Norwich and Norfolk Hospitals Trust, Norwich
  - University Hospitals Dorset, Poole
  - Surrey and Sussex Hospital Trust, Redhill

IPD SHARING:
Plan to Share IPD: Undecided
Subject to constraints in patient consent